CLINICAL TRIAL: NCT04074707
Title: Optimizing Oral Iron Supplementation Regimens During Pregnancy Using Serum Hepcidin Profiles and Iron Stable Isotopes: Defining a Dosing Regimen With Maximal Absorption and Minimal Gastrointestinal Side Effects
Brief Title: Defining a Dosing Regimen With Maximal Absorption for Oral Iron Supplementation During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof.Dr., Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TIPS
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Iron Deficiency Anemia of Pregnancy
MeSH Terms: interventions — ferrous fumarate

STUDY DESIGN:
Intervention Model Description: each subject acts as her own control by going through all the three supplementation cycles. Women will be randomly assigned to start with the 60mg daily vs alternate day, 120mg daily vs alternate day or 120mg daily vs every third day supplementation cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oral iron supplementation (Experimental): Participants go through 3 cycles of oral iron Supplementation (60mg daily vs alternate day dosing, 120mg daily vs alternate day dosing, 120mg daily vs every third-day dosing)
  Interventions: Dietary Supplement: Labeled iron solution (60mg and 120mg Ferrous Fumarate)

INTERVENTIONS:
Dietary Supplement: Labeled iron solution (60mg and 120mg Ferrous Fumarate) — 3 doses of 60mg iron as ferrous fumarate are given on one consecutive day and one alternate day (e.g., days 1, 2, 4); 3 doses of 120mg iron as ferrous fumarate are given on one consecutive and one alternate day (e.g., days 20, 21, 23); 3 doses of 120mg iron as ferrous fumarate are given on one consecutive and one 3rd day (e.g., days 37, 38, 41). Iron doses are labeled with 4mg of a stable isotope in 200ml deionized water (57Fe, 58Fe or 54Fe). Participants will be randomly assigned to start with 60mg iron daily vs alternate day dosing, 120mg daily vs alternate day dosing or 120mg daily vs every-third day dosing.

SUMMARY:
Iron deficiency anemia (IDA) is common during pregnancy and has adverse effects on the mother, fetus and newborn. Oral iron supplements are usually recommended to prevent ID/IDA during pregnancy.

The aim of this study is to define an iron supplementation schedule with maximal absorption using serum hepcidin profiles and stable iron isotopes in pregnant women. In this randomized, open-label trial, fractional and total iron absorption will be compared from daily dosing with 60 mg iron versus alternate day and every third day dosing with 120 mg iron in pregnant Thai women with low iron stores (n=28) during their second trimester of pregnancy.

This study could have wide impact, providing the evidence base for revised, improved recommendations for iron supplementation during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* gestational week 14-16 at study start
* singleton pregnancy
* Serum ferritin SF <60 µg/L
* non-anemic or mildly anemic, defined as hemoglobin (Hb) >10 g/dL
* female aged 18-45 years
* healthy Thai woman

Exclusion Criteria:

* acute or chronic disease
* taking medications that could influence iron absorption
* smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 30 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption in % | Day 18
  Erythrocyte incorporation of stable iron isotopes 14 days after the last supplement intake of the 60mg daily vs alternate day cycle
Fractional iron absorption in % | Day 35
  Erythrocyte incorporation of stable iron isotopes 14 days after the last supplement intake of the 120mg daily vs alternate day cycle
Fractional iron absorption in % | Day 53
  Erythrocyte incorporation of stable iron isotopes 14 days after the last supplement intake of the 120mg daily vs every third day cycle
Total iron absorption in % | Day 18
  Fractional iron absorption measured from the 60mg daily vs alternate day cycle multiplied by the dose
Total iron absorption in % | Day 35
  Fractional iron absorption measured from the 120mg daily vs alternate day cycle multiplied by the dose
Total iron absorption in % | Day 53
  Fractional iron absorption measured from the 120mg daily vs every third day cycle multiplied by the dose
Serum Hepcidin | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
Serum Hepcidin | Day 2
  in the morning before second supplement intake of the 60mg daily vs alternate day cycle
Serum Hepcidin | Day 4
  in the morning before third supplement intake of the 60mg daily vs alternate day cycle
Serum Hepcidin | Day 18
  in the morning before first supplement intake of 120mg daily vs alternate day cycle
Serum Hepcidin | Day 19
  in the morning before second supplement intake of 120mg daily vs alternate day cycle
Serum Hepcidin | Day 21
  in the morning before third supplement intake of 120mg daily vs alternate day cycle
Serum Hepcidin | Day 35
  in the morning before first supplement intake of the 120mg daily vs every third day cycle
Serum Hepcidin | Day 36
  in the morning before second supplement intake of the 120mg daily vs every third day cycle
Serum Hepcidin | Day 39
  in the morning before third supplement intake of the 120mg daily vs every third day cycle
Serum Hepcidin | Day 53
  in the morning 14 days after last supplement intake the 120mg daily vs every third day cycle

SECONDARY OUTCOMES:
Serum Ferritin (SF) | Screening
  in the morning before first supplement intake
Serum Ferritin (SF) | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
Serum Ferritin (SF) | Day 18
  in the morning before first supplement intake of the 120mg daily vs alternate day cycle
Serum Ferritin (SF) | Day 35
  in the morning before first supplement intake of the 120mg daily vs every third day cycle
Serum Ferritin (SF) | Day 53
  in the morning 14 days after last supplement intake of the 120mg daily vs every third day cycle
Hemoglobin (Hb) | Screening
  in the morning before first supplement intake
Hemoglobin (Hb) | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
Hemoglobin (Hb) | Day 18
  in the morning before first supplement intake of the 120mg daily vs alternate day cycle
Hemoglobin (Hb) | Day 35
  in the morning before first supplement intake of the 120mg daily vs every third day cycle
Hemoglobin (Hb) | Day 53
  in the morning 14 days after last supplement intake of the 120mg daily vs every third day cycle
Soluble transferrin receptor (sTfR) | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
Soluble transferrin receptor (sTfR) | Day 18
  in the morning before first supplement intake of the 120mg daily vs alternate day cycle
Soluble transferrin receptor (sTfR) | Day 35
  in the morning before first supplement intake of the 120mg daily vs every third day cycle
Soluble transferrin receptor (sTfR) | Day 53
  in the morning 14 days after last supplement intake of the 120mg daily vs every third day cycle
C-reactive protein (CRP) | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
C-reactive protein (CRP) | Day 18
  in the morning before first supplement intake of the 120mg daily vs alternate day cycle
C-reactive protein (CRP) | Day 35
  in the morning before first supplement intake of the 120mg daily vs every third day cycle
C-reactive protein (CRP) | Day 53
  in the morning 14 days after last supplement intake of the 120mg daily vs every third day cycle
Alpha-1-acid glycoprotein (AGP) | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
Alpha-1-acid glycoprotein (AGP) | Day 18
  in the morning before first supplement intake of the 120mg daily vs alternate day cycle
Alpha-1-acid glycoprotein (AGP) | Day 35
  in the morning before first supplement intake of the 120mg daily vs every third day cycle
Alpha-1-acid glycoprotein (AGP) | Day 53
  in the morning 14 days after last supplement intake of the 120mg daily vs every third day cycle
Serum Hepcidin | Day 1
  in the afternoon after first supplement intake of the 60mg daily vs alternate day cycle
Serum Hepcidin | Day 18
  in the afternoon after first supplement intake of the 120mg daily vs alternate day cycle
Serum Hepcidin | Day 53
  in the afternoon 14 days after third supplement intake of the 120mg daily vs every third day cycle
Serum Iron (SFe) | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
Serum Iron (SFe) | Day 2
  in the morning before second supplement intake of the 60mg daily vs alternate day cycle
Serum Iron (SFe) | Day 4
  in the morning before third supplement intake of the 60mg daily vs alternate day cycle
Serum Iron (SFe) | Day 1
  in the afternoon after first supplement intake of the 60mg daily vs alternate day cycle
Serum Iron (SFe) | Day 18
  in the morning before the first supplement intake of the 120mg daily vs alternate day cycle
Serum Iron (SFe) | Day 19
  in the morning before the second supplement intake of the 120mg daily vs alternate day cycle
Serum Iron (SFe) | Day 21
  in the morning before the third supplement intake of the 120mg daily vs alternate day cycle
Serum Iron (SFe) | Day 18
  in the afternoon after the first supplement intake of the 120mg daily vs alternate day cycle
Serum Iron (SFe) | Day 35
  in the morning before the first supplement intake of the 120mg daily vs every third day cycle
Serum Iron (SFe) | Day 36
  in the morning before the second supplement intake of the 120mg daily vs every third day cycle
Serum Iron (SFe) | Day 39
  in the morning before the third supplement intake of the 120mg daily vs every third day cycle
Serum Iron (SFe) | Day 53
  in the morning 14 days after the last supplement intake of the 120mg daily vs every third day cycle
Serum Iron (SFe) | Day 53
  in the afternoon 14 days after the last supplement intake of the 120mg daily vs every third day cycle
Total Iron Binding Capacity (TIBC) | Day 1
  in the morning before first supplement intake of the 60mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 2
  in the morning before second supplement intake of the 60mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 4
  in the morning before third supplement intake of the 60mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 1
  in the afternoon after first supplement intake of the 60mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 18
  in the morning before first supplement intake of the 120mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 19
  in the morning before second supplement intake of the 120mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 21
  in the morning before third supplement intake of the 120mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 18
  in the afternoon after first supplement intake of the 120mg daily vs alternate day cycle
Total Iron Binding Capacity (TIBC) | Day 35
  in the morning before first supplement intake of the 120mg daily vs every third day cycle
Total Iron Binding Capacity (TIBC) | Day 36
  in the morning before second supplement intake of the 120mg daily vs every third day cycle
Total Iron Binding Capacity (TIBC) | Day 39
  in the morning before third supplement intake of the 120mg daily vs every third day cycle
Total Iron Binding Capacity (TIBC) | Day 53
  in the morning 14 after last supplement intake of the 120mg daily vs every third day cycle
Total Iron Binding Capacity (TIBC) | Day 53
  in the afternoon 14 after last supplement intake of the 120mg daily vs every third day cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Siebenthal HK, Moretti D, Zimmermann MB, Stoffel NU. Effect of dietary factors and time of day on iron absorption from oral iron supplements in iron deficient women. Am J Hematol. 2023 Sep;98(9):1356-1363. doi: 10.1002/ajh.26987. Epub 2023 Jun 26. PMID 37357807